CLINICAL TRIAL: NCT06093126
Title: Lemborexant for Insomnia in a Patient With Dementia: An N-of-1 Trial
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Shanna Trenaman, Dr., Nova Scotia Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LembN01
Record Dates: First submitted 2023-10-06; First posted 2023-10-23 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Insomnia; Dementia; Frontotemporal Dementia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Dementia; Frontotemporal Dementia | interventions — lemborexant

STUDY DESIGN:
Intervention Model Description: The study will be an N of 1 trial over 8 weeks were treatment with lemborexant given alternated with a placebo in an "ABBABAAB" format.
Masking Description: The subject will not be aware what the treatment is.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- lemborexant (Experimental): The study will be an N of 1 trial over 8 weeks were treatment with lemborexant being alternated with a placebo in an "ABBABAAB" format.
  Interventions: Drug: Lemborexant 5 MG

INTERVENTIONS:
Drug: Lemborexant 5 MG — The participant will receive 8 weeks of treatment Week 1 = placebo Week 2 = lemborexant 5mg Week 3 = lemborexant 10 mg Week 4 = placebo Week 5 = lemborexant 10 mg Week 6 = placebo Week 7 = placebo Week 8 = lemborexant 10 mg
  Other Names: Lemborexant 10 MG

SUMMARY:
Insomnia is a highly common, chronic disorder that is distressful for the patient but also for caregivers and can give rise to a heavy burden on the healthcare team. Sleeping aids like benzodiazepines and other sedatives (e.g., zolpidem, zopiclone) have been widely used to help treat insomnia. However, sleeping aids are also known to cause adverse drug reactions such as drowsiness and dizziness, that increases the risk of falls, driving impairment, visual impairment, cognitive impairment, and upon discontinuation may cause paradoxical rebound insomnia, delirium, and nightmares all of which exacerbate the initial insomnia. All of the negative aspects of sleeping aid use are exaggerated for older, frail adults.

Some patients experience an early (young-age) onset dementia with a substantial component of insomnia. Due to the many risks associated with traditional sleeping aids they are often inappropriate in adults living with cognitive impairment and/or frailty. Lemborexant comes from a new class of medications for insomnia. Lemborexant is a dual orexin receptor antagonist that blocks the binding of wake-promoting neuropeptides orexin A and orexin B to their receptors orexin 1 receptor (OX1R) and orexin 2 receptor (OX2R), which is thought to suppress wake drive. Unlike other traditional sleeping aids, lemborexant has not shown to be significantly associated with driving impairment, rebound insomnia, or dependence/withdrawal symptoms. Also, in clinical trials it only rarely causes the types of adverse events associated with benzodiazepines and other traditional sedatives and is less often associated with discontinuations due to adverse events.

While lemborexant is available on the Canadian market it is unclear how this medication will be tolerated by patients living with an early onset dementia. Understanding the effectiveness and tolerability of lemborexant will be helpful in an N of 1 trial to understand the details of effect and effectiveness in individual patients.

DETAILED DESCRIPTION:
Background & Rationale Insomnia is a highly common, chronic disorder that is distressful for the patient but also for caregivers and can give rise to a heavy burden on the healthcare team. Sleeping aids like benzodiazepines and other sedatives (e.g., zolpidem, zopiclone) have been widely used to help treat insomnia. However, sleeping aids are also known to cause adverse drug reactions such as drowsiness and dizziness, that increases the risk of falls, driving impairment, visual impairment, cognitive impairment, and upon discontinuation may cause paradoxical rebound insomnia, delirium, and nightmares all of which exacerbate the initial insomnia. All of the negative aspects of sleeping aid use are exaggerated for older, frail adults.

Some patients experience an early (young-age) onset dementia with a substantial component of insomnia. Due to the many risks associated with traditional sleeping aids they are often inappropriate in adults living with cognitive impairment and/or frailty. Lemborexant comes from a new class of medications for insomnia. Lemborexant is a dual orexin receptor antagonist that blocks the binding of wake-promoting neuropeptides orexin A and orexin B to their receptors orexin 1 receptor (OX1R) and orexin 2 receptor (OX2R), which is thought to suppress wake drive. Unlike other traditional sleeping aids, lemborexant has not shown to be significantly associated with driving impairment, rebound insomnia, or dependence/withdrawal symptoms. Also, in clinical trials it only rarely causes the types of adverse events associated with benzodiazepines and other traditional sedatives and is less often associated with discontinuations due to adverse events.

While lemborexant is available on the Canadian market it is unclear how this medication will be tolerated by patients living with an early onset dementia. Understanding the effectiveness, tolerability, and safety of lemborexant will be helpful in an N of 1 trial to understand the details of effect and effectiveness in individual patients living with dementia and insomnia.

Hypothesis The investigators hypothesize that lemborexant will be effective and safe in the treatment of insomnia in adults living with both early-onset dementia and concomitant sleep difficulty.

Objective The objective of this study is to evaluate lemborexant for efficacy and safety as a sedative medication for insomnia in adults living with both early-onset dementia and insomnia.

Methods This is an investigator led N of 1 trial for adults with early onset dementia and insomnia. While this trial is designed for a particular patient case the investigators anticipate that there may be opportunities in the future for this N of 1 trial to be redeployed additional times to other adults living with early onset dementia.

Study Procedures:

1. Patients identified to have early onset dementia and insomnia by a co-principal investigator during routine patient care will be considered for the N of 1 trial.
2. The other co-investigator will then meet the potential patient, review of the project details and study objectives. There will be a discussion of risks and benefits and the consent form will be reviewed. There will be an invitation for the patient to provide informed consent. Given that the study will include people living with dementia and cognitive impairment investigators will ensure that a caregiver or substitute decision maker will participate in these discussions as well.
3. Once the patient provides informed consent with support from a substitute decision maker if necessary, the patient will be considered enrolled in the study and will be provided with (1) Study medication and (2) Study reporting tool.

(1) Study medication will be provided for an 8 week period. Medications will be dispensed in an ABiBABAAB sequence where each letter represents 7 days of treatment, A represents placebo, Bi represents lemborexant 5mg and B represents lemborexant 10 mg. This doubly counterbalanced design to defends against both linear secular trends and nonlinear trends. Medication will be provided in 7 day packs (plastic or cardboard dosette) marked to correspond to the assigned treatment week and assigned as follows.

Week 1 = placebo Week 2 = lemborexant 5mg Week 3 = lemborexant 10 mg Week 4 = placebo Week 5 = lemborexant 10 mg Week 6 = placebo Week 7 = placebo Week 8 = lemborexant 10 mg Medications will be placed inside an opaque capsule to minimize the difference in appearance for the active and inactive treatments. Dispensing details of the 3 treatments will be provided with each of the 8 week long medication supplies. Please note that there will be no washout time between treatment periods (For practical purposes, washout periods may not be necessary when treatment effects (e.g., therapeutic half-lives) are short relative to the length of the treatment periods. Since treatment half-lives are often not well characterized and vary among individuals, the safest course may be to choose treatment lengths long enough to accommodate patients with longer than average treatment half-lives and to take frequent (e.g., daily) outcome measurements.

(2) The patient will also be provided with a Study reporting tool (Appendix 1) where they can record details of drug response and any other noticed events/effects.

4. The participant/caregiver will receive weekly follow up phone calls by the researcher to report the efficacy and harms that the participant experienced in the last 7 days for the 8-week duration and ensure that the treatment is being tolerated. These details will be recorded for consideration and assessment when determining patient response.

5. Efficacy outcome that will be measured in the Study Reporting tool will include: i) total sleep time, ii) sleep onset latency (SOL), iii) wake time after sleep onset (WASO), iv) sleep efficiency, v) number of awakenings to be measured nightly based on patient and caregiver estimate, vi) quality of sleep (see Appendix 2), vii) quality of life of both the patient and the caregiver.

Risk outcome that will be measured will include:

i) presence & severity of adverse drug reactions (ADRs) (somnolence, headache, sleep paralysis, etc.), ii) patient's willingness to drop-out due to ADRs. Furthermore, provision of follow-up care will be ensured by the co-investigator.

Statistical Analysis N of 1 trials are completed with a signal analysis which analyzes the differences in effect between the periods of treatment and the periods of comparator. In this study the treatment will be lemborexant and the comparator will be placebo. Investigators will assess each of the efficacy measures and risk outcomes and then compare across periods of active treatment and comparator.

ELIGIBILITY:
Inclusion Criteria:

* Identified by clinician investigator to have early-onset dementia and a significant component of insomnia.

Exclusion Criteria:

* Known sleep disorders that are contraindications for orexin antagonist therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2028-12-11 (Estimated); Study Completion 2028-12-11 (Estimated)

PRIMARY OUTCOMES:
Total sleep time | Daily for 8 weeks
  Total number of hours of sleep
Sleep onset latency (SOL) | Daily for 8 weeks
  How long it takes to fall asleep the first time the patient goes to sleep in minutes
Wake time after sleep onset | Daily for 8 weeks
  How long the patient is awake overnight
Number of night awakenings | Daily for 8 weeks
  How many times the patient wakes overnight
Quality of sleep | Weekly for 8 weeks
  Based on sleep quality questionnaire

SECONDARY OUTCOMES:
Presence & severity of ADRs | Daily for 8 weeks
  Monitor events that may be related to medication use
Drop-out due to ADR | Daily for 8 weeks
  Monitor events that may be related to medication use

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Scotia Health, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
Not applicable. No planned sharing of results but upon reasonable request findings may be shared if other researchers wish to pursue inclusion as part of the study team and submit ethics approval for that permission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT06093126/Prot_SAP_000.pdf